CLINICAL TRIAL: NCT00037271
Title: Genome Scan for Obesity in a Multi-Ethnic Sample
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1158; R03HL065702 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To scan the genome for obesity in a multi-ethnic sample.

DETAILED DESCRIPTION:
BACKGROUND:

Despite intensive efforts the genetic basis of obesity has been difficult to establish. Linkage analysis using a genome-wide scan can potentially identify genomic regions not previously thought to be associated with susceptibility to obesity and provides a comprehensive test of the consistency of previous studies. The study used the considerable resources generated by the four cooperating networks in the NHLBI-supported "Family Blood Pressure Program" (FBPP) to conduct a genome-wide scan data for obesity.

DESIGN NARRATIVE:

In the Family Blood Pressure Program, microsatellite markers were typed at a density of -10cM by the Mammalian Genotyping Service (MGS) in Marshfield, WI. The complete data set was to include 9,940 individuals representing 4 ethnic groups (white, black, Hispanic and Asian). Obesity was characterized as a weight/height ratio (body mass index) and waist/hip ratio. This data set was larger than any prior genome scan for obesity, and the inclusion of multiple ethnic groups made it possible to examine genetic heterogeneity. The specific aims of the study were to conduct linkage and association analyses to localize regions influencing obesity. Investigators worked closely with the FBPP Coordinating Center (Washington University, St. Louis) and investigators from each of the four FBPP networks. Evidence was sought for consistency between results obtained from analyses of the genome scan performed by each of the individuals, and results summarized from the literature, with those found in meta-analysis.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Study Completion 2003-03 (Actual)

REFERENCES:
- [Background] Zhu X, Cooper RS, Luke A, Chen G, Wu X, Kan D, Chakravarti A, Weder A. A genome-wide scan for obesity in African-Americans. Diabetes. 2002 Feb;51(2):541-4. doi: 10.2337/diabetes.51.2.541. PMID 11812767
- [Background] Zhu X, Zhang S, Zhao H, Cooper RS. Association mapping, using a mixture model for complex traits. Genet Epidemiol. 2002 Aug;23(2):181-96. doi: 10.1002/gepi.210. PMID 12214310
- [Background] Wu X, Cooper RS, Borecki I, Hanis C, Bray M, Lewis CE, Zhu X, Kan D, Luke A, Curb D. A combined analysis of genomewide linkage scans for body mass index from the National Heart, Lung, and Blood Institute Family Blood Pressure Program. Am J Hum Genet. 2002 May;70(5):1247-56. doi: 10.1086/340362. Epub 2002 Mar 28. PMID 11923912
- [Background] Zhu X, Chang YP, Yan D, Weder A, Cooper R, Luke A, Kan D, Chakravarti A. Associations between hypertension and genes in the renin-angiotensin system. Hypertension. 2003 May;41(5):1027-34. doi: 10.1161/01.HYP.0000068681.69874.CB. Epub 2003 Apr 14. PMID 12695419
- [Background] Huang J, Jiang Y. Genetic linkage analysis of a dichotomous trait incorporating a tightly linked quantitative trait in affected sib pairs. Am J Hum Genet. 2003 Apr;72(4):949-60. doi: 10.1086/374568. Epub 2003 Mar 17. PMID 12644967
- [Background] Zhu X, Yan D, Cooper RS, Luke A, Ikeda MA, Chang YP, Weder A, Chakravarti A. Linkage disequilibrium and haplotype diversity in the genes of the renin-angiotensin system: findings from the family blood pressure program. Genome Res. 2003 Feb;13(2):173-81. doi: 10.1101/gr.302003. PMID 12566395
- [Background] Zhu X, Cooper RS. Linkage disequilibrium analysis of the renin-angiotensin system genes. Curr Hypertens Rep. 2003 Feb;5(1):40-6. doi: 10.1007/s11906-003-0009-x. PMID 12530934